CLINICAL TRIAL: NCT02943044
Title: Characterization of Physiological and Morphological Features of Clinical Head & Neck Squamous Cell Carcinomas (HNSCCs) Using a Quantitative Optical Sensor
Brief Title: Quantitative Optical Sensor Findings in Head & Neck Squamous Cell Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zenalux Biomedical, Inc. (Industry)
Collaborators: Duke University (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: Pro00065967; 5R42CA156901-03 (NIH)
Record Dates: First submitted 2016-10-21; First posted 2016-10-24 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Squamous Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Squamous Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: No intervention, this is an observational study — Non interventional, non-invasive measurements of tissue samples suspected of squamous cell carcinoma using an optical probe.

SUMMARY:
The goal of this study is to determine the optical spectroscopy characteristics of tumor in patients with head and neck squamous cell carcinoma (HNSCC). HNSCC constitutes over 90% of all head and neck cancers. These spectroscopy measurements will be compared with pathological diagnosis of tissue biopsies from the same site. These readings will be performed in the operating room during routine endoscopy with biopsy and tumor mapping of patients who have a suspected squamous cell carcinoma of the head and/or neck. Furthermore, a built in pressure sensor will be used to compare biopsy sites with their benign counterparts. If successful, the optical measurements could be used to survey for and delineate the extent of malignancies in a noninvasive manner. This would be especially helpful for clinic visits where suspicious lesions are seen and would otherwise require biopsy for diagnosis. Immediate benefits would include patients with unknown primaries in which numerous directed biopsies are obtained from multiple head and neck sites.

DETAILED DESCRIPTION:
PURPOSE OF THE STUDY:

HYPOTHESES:

Noninvasive optical spectroscopic measurements of Head and Neck Squamous Cell Carcinoma (HNSCC) result in unique signatures that can differentiate between dysplasia, normal, other benign conditions as well as response to radiation therapy as assessed by clinical and histopathological methods.

STUDY OBJECTIVES

1. Characterization of physiological and morphological features of clinical HNSCCs using a spectroscopy based quantitative optical sensor
2. Evaluate the built-in pressure sensor of the probe as a means of making more measurements at a more consistent, narrower pressure range.

This device will be used to compare spectroscopy measurements with histopathological diagnoses. Subjects will undergo optical measurements at the time of routine biopsy for a suspected squamous cell carcinoma of the head and/or neck . Diffuse reflectance spectroscopy measurements from each lesion of clinical interest, as well as distant normal tissue. Three to five repeated scans will be obtained at each measured site. The clinical "tumor" site will then be biopsied. Samples will not be collected from normal tissue for biopsy. The results of the spectroscopy measurements are for research purposes only and will not be used to confirm a subject's diagnosis.

The optical spectrometer does not breach any skin defense barrier. As this study involves noninvasive optical measurements of tissues, no significant safety concerns are anticipated. The protocol measurements take less than one minute per site. The total amount of extended OR time is expected to be less than 5 minutes. No additional charges to the subject and/or insurance company is expected.

Qualitative analysis will be performed to describe whether there is correlation between spectroscopy measurements and pathologic diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing panendoscopy and biopsy for suspected squamous cell carcinoma of the head and neck.
* patient is > 24 to <89 years of age
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* < 24 years of age, >89 years of age
* Unable to provide written informed consent.

Ages: 24 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients between the ages of 24 - 89 who are scheduled for routine panendoscopy and biopsy for suspected Head & Neck Squamous Cell Carcinoma.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2016-12 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Optical spectroscopic measurements of tumors in patients with HNSCC compared to the histopathologic diagnosis. | During the time of routine biopsy, approximately 5 minutes will be used to perform the optical measurements

SECONDARY OUTCOMES:
Optimal pressure levels of the optical probe | During the time of routine biopsy, approximately 5 minutes will be used to perform the optical measurements
Added pressure sensing and self-calibration features of the optical probe improves specificity and sensitivity to differentiate HNSCC from their benign counterparts | During the time of routine biopsy, approximately 5 minutes will be used to perform the optical measurements

CONTACTS AND LOCATIONS:
Overall Officials: Walter Lee, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Data will be de-identified prior to being shared outside of Duke.